CLINICAL TRIAL: NCT02485379
Title: Improvement in the Detection of Aggressive Prostate Cancer by Targeted Biopsies Using Multiparametric MRI Findings
Brief Title: Assessment of Prostate MRI Before Prostate Biopsies
Acronym: MRI-FIRST01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL14_0440
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Multiparametric MRI; Prostate biopsy; Targeted biopsy; Comparative study
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate biopsy (Other): Systematic biopsies (SB) and targeted biopsies (TB) are performed in the same patients by two independent operators. In patients without abnormalities on mp-MRI, no targeted biopsies will be carried out and the detection of "clinically significant cancer" will be considered as negative for the TB strategy.
  Interventions: Procedure: Prostate biopsy

INTERVENTIONS:
Procedure: Prostate biopsy — Systematic biopsies (SB) and targeted biopsies (TB) are performed in the same patients by two independent operators. In patients without abnormalities on mp-MRI, no targeted biopsies will be carried out and the detection of "clinically significant cancer" will be considered as negative for the TB strategy.

SUMMARY:
Background: Prostate cancer is difficult to detect using ultrasound. As a result, in case of suspicion of prostate cancer based on digital rectal examination (DRE) or Prostate Specific Antigen (PSA) level, it is currently recommended to perform "blinded" systematically distributed biopsies with 10-18 samples obtained from predefined locations in the gland.

These so-called systematic biopsies (SB) may lead to improper patient management by (i) missing clinically significant cancer, especially in the anterior half of the gland that tends to be undersampled, (ii) inducing chance detection of clinically insignificant cancer foci that may result in overtreatments, (iii) undersampling the tumor foci and thus underestimating their volume and aggressiveness.

Multiparametric Magnetic Resonance Imaging (mp-MRI) has yielded promising results in detecting aggressive (Gleason ≥7) prostate cancers. Several monocenter studies showed that targeted biopsies (TB) based on mp-MRI findings could detect significantly more aggressive cancers, reduce the diagnosis of clinically insignificant cancers, and better evaluate the aggressiveness of detected cancers than SB. However, these monocenter studies only provide low-level evidence and three recent independent reviews of literature concluded that there was a need for a robust multicenter trial evaluating the diagnostic yield of TB as compared to SB. This is particularly important since many academic and private centers in France already perform mp-MRI before prostate biopsy in daily routine. Therefore the risk is that this approach becomes the norm without being properly evaluated and it is crucial and urgent to perform a controlled multicentric study to provide high-level evidence as to whether mp-MRI should or should not be obtained before prostate biopsy.

One controlled multicentric study has been published recently in which SB and TB had been obtained by two different operators in 95 patients. TB yielded a significantly higher detection rate for all prostate cancers (69% vs 59%, p=0.033) and for clinically significant cancers (67% vs 52%, p=0.0011). However, this study was limited by the fact that patients with negative mp-MRI were not included.

Research hypotheses: There is currently no robust multicenter trial comparing prostate TB based on mp-MRI findings versus the current standard of care (SB). We propose a multicentre prospective trial comparing the results of SB and TB performed in the same patients by two independent operators. Our hypothesis is that TB detects aggressive (Gleason ≥7) cancers in a significantly higher percentage of patients than SB.

Main objective: To compare the percentage of patients with "clinically significant cancer" (using definition A, i.e. cancer with Gleason score ≥7) detected by SB versus TB.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for prostate mp-MRI before a first set of prostate biopsies, with a planned time interval of less than 3 months between MRI and biopsies
* Age ≤75 years
* PSA level ≤20 ng/mL
* Clinical stage ≤T2c
* Patient insured under the French social security system or beneficiary of an equivalent regime

Exclusion Criteria:

* Contraindication to transrectal biopsy
* Contraindication to MRI
* History of hip prosthesis
* History of androgen deprivation therapy
* Patients with history of prostate cancer diagnosed on TURP
* Patients with history of pelvic radiation therapy (whatever the reason)
* Patient deprived of freedom following a court or administrative order
* Patient under guardianship or under legal guardianship

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Detection of "clinically significant cancer" (using definition A, i.e. Gleason ≥7 cancers) in at least one core of SB or TB. | Between 1 and 4 months after the enrollment

SECONDARY OUTCOMES:
To compare the percentage of patients with "clinically significant cancer" (using definition B, i.e. any Gleason ≥7 cancer or Gleason 6 cancer with at least one sample with ≥6 mm of cancer) detected by SB and TB. | Between 1 and 4 months after the enrollment
To compare the percentage of patients with "clinically significant cancer" (using definition C, i.e. any Gleason ≥7 (4+3) cancer) | Between 1 and 4 months after the enrollment
To compare the percentage of patients with "clinically insignificant cancer" (defined as a Gleason ≤6 cancer with ≤2 positive samples and <3 mm of cancer on the positive samples) detected by SB and TB. | Between 1 and 4 months after the enrollment
To compare the percentage of patients with Gleason ≥7 cancer detected by SB and TB in different subgroups | Between 1 and 4 months after the enrollment
  The different subgroups are :
  * Patients with clinical stage T1c (i.e. normal DRE) versus T2a-T2c,
  * Patients with a PSA level <10 ng/mL versus 10-20 ng/mL,
  * Patients with a prostate volume ≤50 cc versus >50 cc,
  * Patients in whom TB have been performed with ultrasound/MRI fusion versus cognitive guidance
To compare the percentage of patients detected by TB and by SB+TB with "clinically significant cancer" (using definitions A, B and C) and "clinically insignificant" cancer. | Between 1 and 4 months after the enrollment
To compare the percentage of patients with "clinically significant cancer" (using definitions A, B and C) detected by the 2 optional US-guided biopsies and by the regular 12 systematic biopsies. | Between 1 and 4 months after the enrollment
To evaluate the percentage of patients with overall cancer and with "clinically significant cancer" (using definitions A, B and C) on SB and who had a negative MRI | Between 1 and 4 months after the enrollment
To evaluate the percentage of patients with overall cancer and "clinically significant cancer" (using definitions A, B and C) on SB and who had a positive MRI in the sextant(s) that were positive on SB. | Between 1 and 4 months after the enrollment
To evaluate the percentage of patients with discordant results (Gleason score, maximum length of invasion) between the local pathological analysis and between the central pathological review. | Between 1 and 4 months after the enrollment

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Groupe Hospitalier Pellegrin - CHU de Bordeaux, Bordeaux
  - Hôpital Michallon - CHU de Grenoble, Grenoble
  - Hôpital Huriez - CHU de Lille, Lille
  - Hôpital Privé La Louvière, Lille
  - CLIMAL (Centre Libéral Imagerie Médicale Agglomération Lille), Lille
  - Centre Hospitalier St Joseph St Luc, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - Clinique Jules Verne, Nantes
  - Hopital Pitie Salpetriere, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne, Saint-Etienne
  - Clinique Urologique Nantes Atlantis, Saint-Herblain
  - IRMAS, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil - CHU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole - CHU de Toulouse, Toulouse
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Rouviere O, Puech P, Renard-Penna R, Claudon M, Roy C, Mege-Lechevallier F, Decaussin-Petrucci M, Dubreuil-Chambardel M, Magaud L, Remontet L, Ruffion A, Colombel M, Crouzet S, Schott AM, Lemaitre L, Rabilloud M, Grenier N; MRI-FIRST Investigators. Use of prostate systematic and targeted biopsy on the basis of multiparametric MRI in biopsy-naive patients (MRI-FIRST): a prospective, multicentre, paired diagnostic study. Lancet Oncol. 2019 Jan;20(1):100-109. doi: 10.1016/S1470-2045(18)30569-2. Epub 2018 Nov 21. PMID 30470502